CLINICAL TRIAL: NCT00444002
Title: Hepatitis C Infection With Liver Steatosis Compared to Hepatitis C Infection Without Liver Steatosis: Is There a Difference in Lipid Peroxidation and Indicators of Inflammation?
Brief Title: Oxidative Stress and Fatty Acids in Hepatitis C
Status: Completed | Type: Observational
Sponsor: Johane Allard (Other)
Collaborators: Canadian Association of Gastroenterology (Industry)
Responsible Party: Sponsor-Investigator, Johane Allard, Prof. Dr., University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Other Study IDs: 05-0305 AE
Record Dates: First submitted 2007-03-06; First posted 2007-03-07 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Hepatitis C; Hepatic Steatosis
Keywords: Hepatitis C; Steatosis; Oxidative Stress; Antioxidants; Inflammation; Fatty acids
MeSH Terms: conditions — Hepatitis C; Fatty Liver; Inflammation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hepatitis C - Steatosis: Patients with chronic Hep C infection undergoing liver biopsy with >=5% steatosis on liver biopsy
- Hepatitis C - no steatosis: Patients with chronic Hep C infection without steatosis on liver biopsy (<5% of hepatocytes involved)

SUMMARY:
Hepatitis C virus infection (HCV) is a major health concern in Canada and worldwide. Chronic HCV can cause progressive liver damage leading to inflammation, scarring and, in some cases, cirrhosis or liver cancer. It has been shown that fat accumulation in the liver can accelerate the disease progression and is therefore a risk factor in HCV patients.

However, the exact mechanism(s) by which fat accumulation in the liver is involved in disease progression are not clear yet. It is possible that the presence of fat provides a liver susceptible to a second injurious process which leads to scarring. Candidates for this second "hit" may include insulin resistance, leading to accumulation of fat within the liver cells and secondly oxidation of these lipids. In turn, lipid peroxidation can lead to production of reactive oxygen species (unstable molecules that can damage cells) and cytokines (signal molecules that promote inflammation) resulting in more oxidative stress and liver damage.

Aim of the study is to find out, whether patients with HCV and fatty liver have increased oxidative stress and inflammation than patients with HCV without fatty liver, and whether this is associated with a different nutritional status.

DETAILED DESCRIPTION:
Hypothesis: Patients with Hepatitis C and steatosis are more oxidatively stressed than those without steatosis. This is associated with 1) increased liver lipid peroxides and cytokines (TNF-alpha, TGF-beta); 2) altered unsaturated fat status (intake, tissue storage as measured in red blood cells); 3) reduced antioxidant status.

Objectives: To assess oxidative stress and nutritional status in patients with Hepatitis C and steatosis on liver biopsy and to compare the results to the same parameters measured in patients with Hepatitis C and no steatosis.

Measurements:

Primary outcome: Liver lipid peroxides (LPO)

Secondary outcomes:

Liver: TNF-alpha; liver pathology and immunohistochemistry for adducts of malondialdehyde (MDA), a product of lipid peroxidation (LP), alpha-smooth muscle actin (alpha-SMA), a marker of hepatic stellate cell activation; and transforming growth factor (TGF-beta), a profibrogenic cytokine involved in fibrogenesis, liver fatty acid composition (substrate for lipid peroxidation).

Oxidative stress and nutrition: Plasma lipid peroxides, plasma antioxidant vitamins, antioxidant status and power, and red blood cell fatty acid composition, 7 day food record, anthropometry.

Other measurements:

Insulin resistance parameters such as blood glucose, insulin, c-peptide, hemoglobin A1c (HbA1c) Blood lipid profile, liver enzymes (as part of standard medical assessment) Subject demographics and medical history will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, age >18 y
* Established hepatitis C infection as confirmed by positive serology and positive hepatitis C RNA in serum
* Convincing evidence of negligible alcohol consumption (<20g of ethanol per day) obtained from a detailed history, confirmed by at least one close relative
* Absence of any other possible cause for liver dysfunction.
* Undergoing routing liver biopsy (usually pre-treatment)

Exclusion Criteria:

* Findings highly suggestive of liver disease of other etiology (e.g. other viral hepatitis, auto-immune chronic hepatitis, primary biliary cirrhosis and genetic liver diseases such as hemochromatosis, alpha-1 antitrypsin deficiency, Wilsons disease and biliary obstruction)
* Anticipated need for liver transplantation in one year or complications of liver disease such as recurrent variceal bleeding, spontaneous porto- systemic encephalopathy, resistant ascites or bacterial peritonitis
* Concurrent medical illnesses contraindicating a liver biopsy (history of unexplained bleeding, hemophilia or abnormal coagulation results as per routine laboratory work-up or other reasons judged by the hepatologist to contraindicate a percutaneous liver biopsy)
* Medications known to precipitate steatohepatitis (corticosteroids, high dose estrogens, methotrexate, amiodarone, calcium channel blockers, sulfasalazine or cloxacillin) in the 6 months prior to entry
* Antioxidant vitamin or n-3 supplementation, ursodeoxycholic acid or any other experimental drug in the 6 months prior to study entry
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic Hep C infection undergoing routine pre-treatment liver biopsy
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2005-07; Primary Completion 2008-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Lipid peroxidation (LPO) in the liver | Single time point
  LPO by commercially available kit

SECONDARY OUTCOMES:
Hepatic fatty acid composition | Single time point
  Fatty acid and lipid composition measured by gas chromatography and mass spectrometry
Antioxidant power in the liver | Single time point
  Antioxidant power (AOP) measured by test kit
Plasma vitamin C | Single time point
  Plasma vitamin C by colorimetric assay
Tocopherols in plasma | Single time point
  alpha- and gamma-tocopherol in plasma by gas chromatography

OTHER OUTCOMES:
Insulin resistance | Single time point
  Homeostasis model assessment of insulin resistance
Dietary intake | single time point
  Macro- and micronutrient intake by 3-day food protocols

CONTACTS AND LOCATIONS:
Overall Officials: Johane P Allard, MD, FRCPC, Principal Investigator — University Health Network, Toronto General Hospital
Locations (1):
- University Health Network (Toronto General Hospital & Toronto Western Hospital), Toronto, Ontario, Canada

REFERENCES:
- [Result] Arendt BM, Mohammed SS, Aghdassi E, Prayitno NR, Ma DW, Nguyen A, Guindi M, Sherman M, Heathcote EJ, Allard JP. Hepatic fatty acid composition differs between chronic hepatitis C patients with and without steatosis. J Nutr. 2009 Apr;139(4):691-5. doi: 10.3945/jn.108.101782. Epub 2009 Feb 11. PMID 19211827